CLINICAL TRIAL: NCT02184169
Title: Oxygen Consumption-based Assessments of Hemodynamics in Neonates Following Congenital Heart Surgery (Oxy-CAHN Study)
Acronym: Oxy-CAHN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, John Kheir, PI, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00006630
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Transposition of the Great Vessels; Hypoplastic Left Heart Syndrome; Oxygen Consumption Based Assessment of Hemodynamics
Keywords: hemodynamics; neonatal; cardiac disease; congenital heart disease; volumetric oxygen consumption
MeSH Terms: conditions — Transposition of Great Vessels; Hypoplastic Left Heart Syndrome; Heart Diseases; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HLHS (Experimental): Patients undergoing palliative repair.
  Interventions: Device: General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments; Device: Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr
- TGA (Active Comparator): Surgical repair of TGA.
  Interventions: Device: General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments; Device: Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr

INTERVENTIONS:
Device: General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments — Breath to breath VO2 measurements
Device: Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr — Edwards continuous SVO2 measurement system

SUMMARY:
The purpose of the Oxy-CAHN study is to improve the monitoring capabilities of newborn infants recovering from congenital heart surgery. Currently, we utilize important but unsophisticated measures, such as vital signs and lactate measurements, to monitor these patients. Although they are useful in categorizing patients as well or unwell, these signs currently lack the power quantify a patient's risk for cardiac arrest. More to the point, they are mostly indirect measures of what we really are assessing, which is tissue oxygen delivery.

Our group has signiﬁcant expertise with devices which quantify the amount of oxygen that a baby consumes every minute. Historically, these values are more commonly used in combination with other measures to assess nutritional and metabolism status. In critically ill patients, however, the volume of oxygen consumed by a patient may be limited by the amount of oxygen their circulation delivers. This may represent a critical relationship, which has been previously described, but not exploited for the purpose of identifying patients with critically low oxygen delivery.

The aims of this study are therefore (1) to demonstrate that oxygen consumption can be safely and precisely measured continuously in newborns undergoing one of two common congenital heart surgeries, (2) to determine whether postoperative circulatory failure is associated with a precedent change in oxygen consumption, and (3) to determine whether the addition of the oxygen-based measurements (including oxygen consumption and venous oxygen saturations) to standardly measured parameters will add power in predicting which patients will experience postoperative circulatory failure.

If successful, this study may improve our capacity to non-invasively and continuously monitor patients following the highest risk congenital heart surgeries, and in the future,to create an algorithm which quantiﬁes a patients risk for having a cardiac arrest. This may permit providers to intervene on these patients earlier, improving the morbidity and mortality associated with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from birth to 6 months of age
2. HLHS AND no prior operations AND planned S1P or HPOR d-TGA/IVS AND planned ASO
3. Written parental informed consent

Exclusion Criteria:

1. Weight < 2 kg
2. Disease speciﬁc A. HLHS patients: Infants whose surgical plan includes a neonatal biventricularrepair will be excluded.

   B. d-TGA/IVS patients: Newborns with any additional cardiac defect other than an atrial septal defect will be excluded.
3. Patients on ECMO preoperatively
4. Clinically signiﬁcant tracheo-esophageal ﬁstula or known preoperative air leak

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kheir, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mills KI, Kaza AK, Walsh BK, Bond HC, Ford M, Wypij D, Thiagarajan RR, Almodovar MC, Quinonez LG, Baird CW, Emani SE, Pigula FA, DiNardo JA, Kheir JN. Phosphodiesterase Inhibitor-Based Vasodilation Improves Oxygen Delivery and Clinical Outcomes Following Stage 1 Palliation. J Am Heart Assoc. 2016 Nov 2;5(11):e003554. doi: 10.1161/JAHA.116.003554. PMID 27806964

RESULTS

PARTICIPANT FLOW:
Groups:
- TGA With/Without VSD: Surgical repair of TGA.
  General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments: Breath to breath VO2 measurements
  Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr: Edwards continuous SVO2 measurement system
Period: Overall Study
Arm/Group | HLHS | TGA With/Without VSD
Started | 21 | 6
Completed | 21 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TGA/IVS: Surgical repair of TGA.
  General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments: Breath to breath VO2 measurements
  Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr: Edwards continuous SVO2 measurement system
- Total: Total of all reporting groups
Arm/Group | HLHS | TGA/IVS | Total
Number analyzed (Participants) | 21 | 6 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 6 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | .1 (.1) | .1 (.1) | .1 (.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 10 | 4 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Region of surgery
  Participants
    United States | 21 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Consumption
Description: Oxygen consumption is the mass of oxygen gas consumed per minute, measured as the difference between oxygen mass inspired versus exhaled per minute.
Time Frame: While mechanically ventilated, up to 14 days
Measure: Mean (Standard Deviation); unit: mL oxygen/min/m^2
Arm/Group | HLHS | TGA With/Without VSD
Number analyzed (Participants) | 21 | 6
mL oxygen/min/m^2 | 72 (12) | 102 (22)

2. Secondary Outcome: Computed Cardiac Index
Description: A calculated estimate of cardiac index/systemic blood flow based on the Fick principle.
Time Frame: While mechanically ventilated, up to 14 days
Population: The average cardiac index was measured for each patient twice per day
Measure: Mean (Standard Deviation); unit: L/min/m2
Groups:
- Hypoplastic Left Heart Syndrome: Patients undergoing palliative repair.
  General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments: Breath to breath VO2 measurements
  Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr: Edwards continuous SVO2 measurement system
- Transposition of the Great Arteries: Surgical repair of TGA.
  General Electric Healthcare E-COVX Gas Monitoring Module for VO2 Measurments: Breath to breath VO2 measurements
  Edwards Continuous SVO2 Catheter and Monitoring System - 4.5 fr: Edwards continuous SVO2 measurement system
Arm/Group | Hypoplastic Left Heart Syndrome | Transposition of the Great Arteries
Number analyzed (Participants) | 21 | 6
L/min/m2 | 1.3 (0.4) | 2.2 (0.6)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | HLHS | TGA/IVS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/6
Other Adverse Events (participants affected / at risk) | 0/21 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02184169/Prot_SAP_000.pdf